CLINICAL TRIAL: NCT06431386
Title: Optimizing the Synergy Between Behavioural Activation Therapy and Esketamine for Resistant Depression
Brief Title: Behavioural Activation Therapy and Esketamine for Resistant Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prematurely due to significant recruitment challenges.
Sponsor: The Royal's Institute of Mental Health Research (Other)
Responsible Party: Principal Investigator, Dr. Jeanne Talbot, Physician Scientist, The Royal's Institute of Mental Health Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 2024002
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Bipolar Disorder
Keywords: Major Depressive Disorder; Esketamine; Psychotherapy; Behavioural Activation; Bipolar Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Bipolar Disorder | interventions — Therapeutics; Esketamine

STUDY DESIGN:
Intervention Model Description: This pilot study is a single-site, parallel-arm, randomized clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Clinical outcome assessments will be performed by raters blind to treatment allocation and not the treating therapist or physician. Ratings will be acquired prior to treatment administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esketamine + Behavioural Activation Therapy (Experimental): Participants randomized to this arm will be administered esketamine treatment as per standard clinical care in conjunction with behavioural activation (BA) therapy. Both treatments will be initiated in Week 1 of the induction phase (first 4 weeks of esketamine treatment).
  Interventions: Behavioral: Behavioural Activation (BA) Therapy; Drug: Esketamine
- Esketamine Alone (Active Comparator): Participants randomized to this arm will be administered esketamine treatment as per standard clinical care and will be offered a course of BA therapy (12 one hour sessions) after their completion of the trial.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Behavioral: Behavioural Activation (BA) Therapy — Participants will receive weekly one-hour BA sessions on a day they are not receiving esketamine, delivered virtually or in person as per participant preference. The aim is for participants to learn to observe the relationship between what they did, felt, and thought and what was happening around them, and to identify conditions which maintained, increased, or weakened maladaptive behaviours. Functional behaviour analysis will be used in problem and behaviour evaluation and in planning and reviewing changes introduced by participants between sessions. Other techniques include self-observation and self-report, elaboration of activity hierarchies, behaviour programming, rehearsal and behavioural modelling, and contingency management. Between-session homework will develop relevant and rewarding routines to offer reinforcement in each participant's environment. Participants will be offered 12 BA sessions in total.
  Arms: Esketamine + Behavioural Activation Therapy
Drug: Esketamine — Participants will receive intranasal esketamine twice weekly during the induction phase (first 4 weeks of treatment). Maintenance treatments are administered once per week or once every two weeks at the discretion of the treating physician for 8 additional weeks, totaling 12 weeks of esketamine treatment. Dosing for esketamine usually starts at 56mg on Day 1, followed by 56 or 84mg doses for subsequent treatments.

SUMMARY:
This is a randomized clinical trial to test the effectiveness of combining a proven psychological intervention called behavioural activation therapy alongside esketamine treatment for treatment resistant major depressive episodes in individuals with major depressive disorder or bipolar disorder. Encouraging participants to practice new behaviours while their mood is improved through esketamine treatment may lead to more lasting recovery from depression.

DETAILED DESCRIPTION:
Depression is the leading cause of disability in the world and current treatments with medication are limited. Over one-third of individuals with major depressive disorder (MDD) and one quarter of individuals with bipolar disorder (BD) do not benefit from traditional pharmacotherapies, leading to treatment-resistant depressive episodes. Individuals with treatment-resistant depressive episodes (defined as a suboptimal response to two or more appropriate trials of antidepressant medication) have a higher burden of illness, higher healthcare utilization, poorer quality of life, worse occupational and social outcomes, and are at greater risk of death. Treatment-resistance may increase an individual's likelihood of engaging in suicidal behaviours and an estimated 30 percent of individuals with treatment-resistant depressive episodes will have a suicide attempt in their lifetime. To address these gaps in treatment, there has been growing interest in the use of intravenous (IV) ketamine as well as its newly marketed stereoisomer, esketamine, which is delivered intranasally.

The discovery of the rapid antidepressant effects of low doses of ketamine has been hailed as a paradigm shift in psychiatry. However, a remaining challenge to address is the temporary nature of its effects. Ketamine induces neuroplasticity-enhancing effects more than conventional medications for depression. There may be the potential to harness this window of neuroplasticity to facilitate more lasting cognitive and/or behavioural changes through psychotherapy. To date, there are no randomized clinical trials of combined treatment with esketamine and psychotherapy for treatment-resistant depressive episodes. Studies to ensure that individuals can maximally benefit from this novel treatment are needed.

The overall goal of this project is to maximize and sustain the beneficial effects of esketamine through combined treatment with behavioural activation (BA) therapy. The central hypothesis is that combined esketamine and BA therapy will elicit larger and faster decrease in depressive symptoms and more improvement in functional recovery compared with esketamine treatment alone.

The specific aims of this research study are as follows:

Aim 1. To determine if there is a larger decrease in depressive symptoms in participants receiving BA concurrent with esketamine treatment compared to participants receiving esketamine alone.

Aim 2. To compare the speed of antidepressant response in participants receiving BA concurrent with esketamine treatment compared to participants receiving esketamine alone.

Aim 3. To assess if participants receiving BA concurrent with esketamine treatment perceive greater improvement in functioning (self-reported depressive symptoms, quality of life, anhedonia, hopelessness, and work and social functioning) compared to participants receiving esketamine alone.

This study is a single-site, parallel-arm, randomized clinical trial investigating the effects of augmenting esketamine treatment with BA therapy, an empirically supported treatment for depression.

Participants will be randomized to one of two groups: 1) concurrent esketamine and BA therapy started from treatment initiation, or 2) esketamine treatment alone.

Esketamine treatment will be offered as treatment as usual. All study participants will be offered a 12 session course of BA therapy, half will be randomized to receive BA concurrently with their esketamine treatment from initiation. Participants randomized to the esketamine treatment alone arm will be offered a full course of BA sessions after week 12 during the maintenance phase of treatment or at the time esketamine treatment ceases, whichever is earlier.

BA therapy will be delivered virtually or in person according to participant preference (mode of administration will be recorded and included in data analysis as appropriate). The aim of BA therapy is to help individuals learn to observe the relationship between what they did, felt, and thought and what was happening around them, and to identify conditions which maintained, increased, or weakened maladaptive behaviours. Functional behaviour analysis will be used in problem and behaviour evaluation and in planning and reviewing changes introduced by participants between sessions. Other techniques include self-observation and self-report, elaboration of activity hierarchies, behaviour programming, rehearsal and behavioural modelling, and contingency management. Between-session homework will develop relevant and rewarding day-to-day routines liable to offer reinforcement in each participant's environment. An independent expert will assess the quality and adherence to BA for the trial.

This will be the first clinical trial to test the concurrent use of esketamine and a behavioural intervention. The efficacy data for esketamine largely comes from randomized controlled trials and thus may not always reflect the clinical reality for individuals who present for treatment in hospital settings. Conducting research with esketamine in a naturalistic academic-hospital setting will inform clinical practice. The goal is to offer esketamine to individuals as part of a comprehensive treatment plan to help them achieve longer-term recovery as opposed to short-lived decrease in clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Ages 18-65
* Participants meeting criteria for major depressive disorder (MDD) or bipolar disorder, depressive episode without psychotic symptoms according to the Diagnostic and Statistical Manual for Mental Disorders (DSM-5).
* Participants who have not responded adequately to at least two separate courses of treatment with different antidepressants, each of adequate dose and duration, in the current moderate to severe depressive episode.

Exclusion Criteria:

* Depression secondary to a stroke, cancer, or other severe medical illnesses.
* Pregnant, lactating or of childbearing potential and unwilling to use an approved method of contraception during the study.
* A history of intracerebral hemorrhage, vascular disease.
* Active psychotic symptoms.
* Current and/or recent history (<12 months) of substance use/dependence (except for caffeine or nicotine) or problematic current alcohol use or dependence as defined by DSM-5 criteria.
* A diagnosis of major neurocognitive disorder or a Montreal Cognitive Assessment (MOCA) score <24.
* Active suicidal intent with the absence of psychotic symptoms is not an exclusion criterion, as this is not atypical in individuals with treatment-resistant, and/or severe depression (safety monitoring will be carried out by research personnel/study psychiatrists).
* Known history of intolerance or hypersensitivity to ketamine.
* Any other condition that, in the opinion of the PI/study investigator(s), would adversely affect the participant's ability to complete the study or its measures.
* The participant must not be receiving psychotherapy treatment outside the clinical trial for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | Baseline to the end of the induction phase (week 4); additional efficacy assessment time points will include end of weeks 2, 8 and 12
  Change in Montgomery-Åsberg Depression Rating Scale (MADRS) score

SECONDARY OUTCOMES:
Speed of therapeutic effects | Induction phase (weeks 1-4)
  Time required to first meet response criteria (≥50% improvement in MADRS scores)
Change in participant perceived functioning | Baseline to end of induction phase (week 4), and the end of weeks 8 and 12
  Change in self-reported depressive symptoms, quality of life, anhedonia, hopelessness, and physical, emotional and social functioning

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Talbot, MD PhD FRCP, Principal Investigator — The Royal's Institute of Mental Health Research
Locations (1):
- The Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada